CLINICAL TRIAL: NCT02261571
Title: A Pilot Study to Estimate the Efficacy of Moxibustion Stimulation at Abdominal Acupoints on Quality of Life in Cancer Patients Under Chemotherapy
Brief Title: Impact on Quality of Life by Moxibustion in Chemotherapy for Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Comprehensive and Integrative Medicine Institute of South Korea (Other)
Responsible Party: Principal Investigator, Hyun jung, Jung, assistant professor, The Comprehensive and Integrative Medicine Institute of South Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CIMI-14-01-08
Record Dates: First submitted 2014-10-02; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxibustion (Experimental): A series of moxibustion sessions within six weeks from baseline with adjuvant chemotherapy.
  Interventions: Other: Moxibustion
- Waiting (No Intervention): Participants who will be allocated to waitlist will receive no moxibustion treatments throughout the 6 weeks while receiving adjuvant chemotherapy

INTERVENTIONS:
Other: Moxibustion — In the moxibustion treatment group, 3 moxibustion, 3 acupoints(CV12, CV8, CV54) will be heated with indirected moxibustion.
  The moxibustion will be removed when the patient feel hotness and require remove them
  Arms: Moxibustion

SUMMARY:
Most cancer patients experience multiple symptoms related to chemotherapy and use CAM (complementary and alternative medicine) as an adjunct to conventional treatment. Moxibustion is traditional Korean medical therapeutic method and uses the heat generated by burning herbal preparations containing Artemisia vulgaris to stimulated acupoint.

Herein, the investigators propose an open-label pilot study investigating the effectiveness of moxibustion stimulation at abdominal acupoint on quality of life in cancer patients under chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic histopathology of cancer
* Performance status of 0-2 on the European Cooperative Oncology Group (ECOG) performance scale.
* Patients on chemotherapy currently have plan to receive chemotherapy for more than 6 weeks.
* Follow-up possible during the clinical trial
* Informed signed consent

Exclusion Criteria:

* Patients with Severe Heart disease and hypertension that is not controlled (systolic blood pressure >160 or Diastolic blood pressure >100)
* Patients with diabetes that is not controlled (FBST >180 or BST>250)
* Patients with abdominal injury or severe ascites can't be received moxibustion therapy on abdomen.
* Hypersensitive section to moxibustion treatment
* Inability to comprehend or express oneself in the Korean language
* An Individual deemed to be ineligible by a physician
* Refusal to participate in this trial or to provide informed consent.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
functional Assessment of Cancer Therapy: General (FACT-G) | change from baseline to 6 weeks

SECONDARY OUTCOMES:
Body mass index | change from baseline to 6 weeks
immune function | change from baseline to 6 weeks
  lymphocyte panel(CD3,4,8,19,26), WBC, Differential count
M.D, Anderson symptom Inventory (MDASI) | change from baseline to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Deagu Hanny University Medical center, Deagu, South Korea

REFERENCES:
- [Background] Lee MS, Kang JW, Ernst E. Does moxibustion work? An overview of systematic reviews. BMC Res Notes. 2010 Nov 5;3:284. doi: 10.1186/1756-0500-3-284. PMID 21054851
- [Background] Lee MS, Choi TY, Park JE, Lee SS, Ernst E. Moxibustion for cancer care: a systematic review and meta-analysis. BMC Cancer. 2010 Apr 7;10:130. doi: 10.1186/1471-2407-10-130. PMID 20374659